CLINICAL TRIAL: NCT04627883
Title: Effect of Inverse Ratio Ventilation During Induction of General Anesthesia on Safe Apnea Time in Obese Patients:A Randomized Controlled Trial
Brief Title: Effect of Inverse Ratio Ventilation During Induction of General Anesthesia on Safe Apnea Time in Obese Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: General Hospital of Ningxia Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2020-718
Record Dates: First submitted 2020-10-11; First posted 2020-11-13 (Actual); Last update posted 2025-02-17 (Actual); Status verified 2020-10

CONDITIONS: Obesity
Keywords: inverse ratio ventilation; safe apnea time
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Intervention Model Description: Parallel Assignment
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group 1:2 (Other): Patients in the control group had noninvasive positive pressure ventilation with inspiratory-to-expiratory (I : E) ratio of 1:2.
  Interventions: Other: Inspiratory-to-expiratory (I : E) ratio of 1:2
- Group 2:1 (Other): Patients in the IRV group had noninvasive positive pressure ventilation with inspiratory-to-expiratory (I : E) ratio of 2:1.
  Interventions: Other: Inspiratory-to-expiratory (I : E) ratio of 2:1

INTERVENTIONS:
Other: Inspiratory-to-expiratory (I : E) ratio of 1:2 — After preoxygenation and induction of anesthesia, noninvasive positive pressure ventilation with inspiratory-to-expiratory (I : E) ratio of 1:2 for 5 min before endotracheal intubation.
  Arms: Group 1:2
Other: Inspiratory-to-expiratory (I : E) ratio of 2:1 — After preoxygenation and induction of anesthesian, noninvasive positive pressure ventilation with inspiratory-to-expiratory (I : E) ratio of 2:1 for 5 min before endotracheal intubation.
  Arms: Group 2:1

SUMMARY:
The purpose of this study is to investigate the clinical application value of inverse ratio ventilation in obese patients during induction of general anesthesia by studying the effect of inverse ratio ventilation on the safe apnea time.

DETAILED DESCRIPTION:
Inverse ratio ventilation(IRV) can produce mean airway pressure(Pmean)similar to external positive end expiratory pressure(Peep) by increasing inspiratory time. Moreover, the increase of Pmean was not accompanied by the further increase of peak airway pressure (Ppeak) and airway plateau pressure (Pplat), while the application of external peep accompanied with the increase of Pplat increased the risk of barotrauma . High level of Peep increased cardiac load and decreased cardiac output. A number of studies have found that the hemodynamic stability of patients can be achieved when IRV regulates the inspiratory / expiratory ratio in an appropriate range (I: E < 2:1). Therefore, the inverse ratio is considered to be superior to Peep in terms of gas exchange and respiratory mechanics.

ELIGIBILITY:
Inclusion Criteria:

* Obese patients, aged 18-65 years, of either gender, ASA grade II-III, body mass index (BMI) > 30 kg / m2, scheduled for general anesthesia under tracheal intubation, signed informed consent.

Exclusion Criteria:

* Patients who need rapid sequence induction (RSI); patients with expected difficult airway; severe chronic respiratory diseases, such as tuberculosis, bronchitis, bronchial asthma and COPD; patients with severe cardiovascular diseases, such as severe ischemic heart disease and pulmonary hypertension; patients with severe cerebrovascular diseases, such as cerebral hemorrhage and cerebral infarction; patients with abnormal basal metabolic rate, such as pregnancy, thyrotoxicosis, pheochromocytoma; and severe stomach reflux disease; patients with abnormal hemoglobin and hematocrit.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2020-08-17 (Actual); Primary Completion 2022-01-01 (Actual); Study Completion 2022-01-01 (Actual)

PRIMARY OUTCOMES:
Safe Apnea Time | The arterial saturation as measured by pulse oximetry remained at or above 93% after endotracheal intubation immediately.
  The safe apnea time was defined as that period of time during which the arterial saturation as measured by pulse oximetry remained at or above 93% .

SECONDARY OUTCOMES:
EtO2 | After 3 minutes of preoxygenation After 5 minutes of noninvasive positive pressure ventilation
  Fractional concentration of oxygen in end-tidal gas
EtO2 | After 3 minutes of noninvasive positive pressure ventilation
  Fractional concentration of oxygen in end-tidal gas
EtO2 | After 5 minutes of noninvasive positive pressure ventilation
  Fractional concentration of oxygen in end-tidal gas

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - General Hospital of Ningxia Medical University, General Hospital of Ningxia Medical University, Ningxia
  - General Hospital of Ningxia Medical University, Yinchuan, Ningxia

IPD SHARING:
Plan to Share IPD: No